CLINICAL TRIAL: NCT06623188
Title: Treatment of Episodic Migraine With AURICular Neuromodulation: a Prospective Randomized, Placebo-controlled Study
Brief Title: Treatment of Episodic Migraine With AURICular Neuromodulation
Acronym: MENAURIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-05
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular neuromodulation (Experimental)
  Interventions: Other: Auricular neuromodulation
- Sham auricular neuromodulation (Sham Comparator)
  Interventions: Other: Sham auricular neuromodulation

INTERVENTIONS:
Other: Auricular neuromodulation — 3 neuromodulation sessions over 12 weeks
  Arms: Auricular neuromodulation
Other: Sham auricular neuromodulation — 3 neuromodulation sessions over 12 weeks
  Arms: Sham auricular neuromodulation

SUMMARY:
Migraine is a ubiquitous pathology affecting approximately 1 billion individuals and being the leading cause of morbidity worldwide before the age of 50. Migraine treatment consists of two main approaches: acute treatment to relieve headache symptoms and preventive treatment to reduce the frequency of migraine attacks by at least 50%. Preventive treatment involves medications such as beta-blockers, antiepileptics, calcium channel blockers, and a new therapeutic class called calcitonin gene-related peptide (CGRP) inhibitors. While traditional treatments have modest efficacy and limited tolerability, CGRP inhibitors have shown better tolerability and superior efficacy. However, their prescription in France is restricted to neurologists and specialized pain evaluation and treatment units. Additionally, the long-term effects of CGRP inhibition on blood pressure control and vascular homeostasis are not fully understood.

In addition to pharmacological preventive treatment, non-pharmacological approaches have emerged, such as auricular neurostimulation. This can be achieved through electrical stimulation of the cymba conchae, considered a non-invasive alternative to invasive vagal stimulation, and has shown benefits in reducing the number of migraine days compared to a placebo. Another approach involves stimulation of specific areas of the entire auricle using techniques borrowed from auriculotherapy (auricular acupuncture).

The objective of the study is to demonstrate that auricular neuromodulation, performed with a laser device, targeted and personalized on selected areas of the auricle, has a beneficial effect on the number of moderate to severe migraine days per month.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≥ Aged ≤ 60 years
* Moderate to severe Migraine for at least one year
* Migraines appeared before the age of 50 and diagnosed according to IHS (international headache society) criteria.
* Therapeutic failure of at least 2 migraine preventive medications
* Frequency of migraine days ≥ 4 per month and < 15 per month

Exclusion Criteria:

* Pathology of the auricle (e.g. epithelioma)
* Patient treated with botulinum toxin for migraine ≤ 2 months
* Patient treated with anti-cgrp for migraine, with last injection less than 3 months ago
* Patient treated with non-invasive auricular stimulation ( TENS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days in the last 4 weeks of treatment, compared with the initial assessment period (4-week pre-treatment observation). | 4 months

SECONDARY OUTCOMES:
Days without headache or migraine | 6 months
Migraine attacks duration | 6 months
Rate of responders, i.e., patients with a 50% reduction in the number of migraine days after treatment compared with the initial assessment | 6 months
Quality of life of patients measured by Study Short Form 36 (SF-36) questionnaire | 6 months
Functional disability due to headache or migraine as measured by MIgraine Disability Assessment (MIDAS) and Headache Impact Test (HIT-6) questionnaires | 6 months
Use of rescue medication | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - BENNANI, Marseille
  - Hôpital Européen Marseille, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagui E, Kereun E, Guillemet G, Faralli H, Perananda G, Bennani M, Berthelier C. Auricular neuromodulation by low level laser therapy versus placebo laser therapy in prophylactic treatment of episodic migraine: a randomized controlled study protocol. BMC Complement Med Ther. 2025 Oct 14;25(1):371. doi: 10.1186/s12906-025-05068-6. PMID 41088062